CLINICAL TRIAL: NCT00457938
Title: Novel Therapies for Metabolic Complications in Patients With Lipodystrophies
Brief Title: Novel Therapies for Metabolic Complications of Lipodystrophies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Takeda (Industry); Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Abhimanyu Garg, Chairman, Division Nutrition and Metabolic Diseases, Professor Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RO1-074959; DK074959
Record Dates: First submitted 2007-04-04; First posted 2007-04-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Insulin Resistance; Hypertriglyceridemia; Diabetes; Hepatic Steatosis
Keywords: lipodystrophy
MeSH Terms: conditions — Insulin Resistance; Hypertriglyceridemia; Diabetes Mellitus; Fatty Liver; Lipodystrophy | interventions — Diet, Fat-Restricted; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low fat diet is the "drug" (Other): Diet 10% fat versus 35% fat
  Interventions: Other: low-fat diet ( Still recruiting ); Other: Diet

INTERVENTIONS:
Other: low-fat diet ( Still recruiting ) — This study will compare 10% fat versus 35% fat diets in terms if effect on liver fat, triglycerides adn other metabolic parameters.
  Other Names: Low fat versus extremely low fat Diet
Other: Diet — 10 % versus 35 % fat in diet

SUMMARY:
Lipodystrophies represent a therapeutic challenge with regards to the management of the diabetes, insulin resistance, hypertriglyceridemia and fatty liver which frequently present in conjunction with significant adipose tissue loss. The purpose of the study and it's four subprojects is to examine the safety and efficacy of various novel interventions designed to improve or resolve the fatty liver, hypertriglyceridemia, and insulin resistance or diabetes that is seen in these patients.

DETAILED DESCRIPTION:
We propose novel therapeutic approaches for the management of metabolic complications in patients with lipodystrophies. The four interventions to be tested are:

Hypothesis 1: An extremely low fat diet.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion criteria:

* Patients with lipodystrophies as diagnosed by clinical criteria
* Any one of the following:

  * Diabetes mellitus, or
  * Fasting serum triglycerides greater than 200 mg/dL, or
  * Fasting serum insulin greater than 30 U/mL, or
  * Hepatic steatosis ( greater than 5.6% hepatic triglyceride content) as demonstrated by 1H MRS.

Exclusion Criteria:

* Known liver disease due to causes other than non-alcoholic steatohepatitis:
* Current alcohol abuse (more than 7 drinks or 210 g per wk for women and more than 14 drinks or 420 g per wk for men).
* Positive serological markers of hepatitis B and C.
* Autoimmune hepatitis, autoimmune cholestatic liver disorders, Wilson disease and Alpha-1-antitrypsin deficiency as indicated by clinical and laboratory tests.
* Drug-induced liver disease
* Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study suggestive of liver cancer.
* Decompensated liver disease as evidenced by clinical features of hepatic failure (variceal bleeding, ascites, hepatic encephalopathy etc.) and laboratory investigations (prolonged prothrombin time, hypoalbuminemia, presence of esophageal varices etc.)
* Use of the drugs which can potentially decrease hepatic steatosis during previous 3 months; high-dose vitamin E, betaine, acetylcysteine, choline and probucol.
* Significant systemic or major illnesses other than liver disease (congestive heart failure, unstable angina, cerebrovascular disease, respiratory failure, renal failure [serum creatinine more then 2 mg/dL], acute pancreatitis, organ transplantation, serious psychiatric disease, and malignancy) that could interfere with the trial and adequate follow up.
* Acute medical illnesses precluding participation in the studies.
* Known HIV infected patient.
* Current substance abuse.
* Pregnant or lactating women.
* Hematocrit of less than 30%.
* History of weight loss ( more than 10%) or use of weight loss drugs such as sibutramine or orlistat in the last 3 months.

Each subproject has additional specific inclusion and exclusion criteria

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Project specific: improvement in serum triglycerides, insulin resistance, liver triglyceride content, liver volume, Hgb A1c, | 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Simha V, Subramanyam L, Szczepaniak L, Quittner C, Adams-Huet B, Snell P, Garg A. Comparison of efficacy and safety of leptin replacement therapy in moderately and severely hypoleptinemic patients with familial partial lipodystrophy of the Dunnigan variety. J Clin Endocrinol Metab. 2012 Mar;97(3):785-92. doi: 10.1210/jc.2011-2229. Epub 2011 Dec 14. PMID 22170723